CLINICAL TRIAL: NCT03734653
Title: Square Wave Testosterone Therapy in Castration Resistant Prostate Cancer
Brief Title: Testosterone Therapy in Castration Resistant Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0821.cc
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Castration-Resistant Prostate Cancer
Keywords: Square Wave Testosterone Therapy; Androgen Deprivation Therapy; Transdermal Testosterone; Feasibility Study
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care; enzalutamide

STUDY DESIGN:
Intervention Model Description: This is a longitudinal pilot, single arm, interventional study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Square Wave Testosterone Therapy + SOC (Experimental): All patients will receive transdermal testosterone. All patients will also receive standard of care enzalutamide. Patients will alternate between the two therapies.
  Interventions: Drug: Transdermal Testosterone; Drug: Standard of Care, Enzalutamide

INTERVENTIONS:
Drug: Transdermal Testosterone — Patients will be prescribed 2 packets of testosterone gel 1% containing 50mg per packet to apply transdermally daily.
Drug: Standard of Care, Enzalutamide — Patients will take four 40mg capsules of enzalutamide for a total daily dose of 160mg.

SUMMARY:
This is an open-labeled, single-arm, interventional pilot study. It is being done to determine the feasibility of the administration of transdermal testosterone alternating with enzalutamide, as well as the safety and efficacy.

DETAILED DESCRIPTION:
The primary endpoint of this trial is to determine the feasibility of the administration of transdermal testosterone alternating with enzalutamide. High dose testosterone has shown activity in phase II studies of patients with castration resistant metastatic prostate cancer; however, these studies have generally employed the intramuscular formulation. It has been hypothesized that the transdermal formulation will show activity but will have less potential for toxicity due to extremely high levels of circulating testosterone (i.e. thrombotic events). In addition, this will allow for a steady state of elevated testosterone, rather than the peaks and troughs seen with the IM approach.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form
2. Male and age > or = 18 years old
3. Stated willingness to comply with all study procedures and be available for the duration of the study
4. Histologically or cytologically proven adenocarcinoma of the prostate
5. Ongoing ADT for prostate cancer with a GnRH analogue/antagonist or bilateral orchiectomy for at least 6 months prior to day 1
6. Patients on a first generation anti-androgen (e.g. bicalutamide, flutamide, nilutamide) must have at least a 6-week washout prior to randomization and must show continued PSA progression
7. Serum testosterone level <50ng/dL at the screening visit
8. Progressive disease at screening as defined by one or more of the following criteria:

   * PSA progression: minimum of 2 rising values within an interval of >1 week between values. And a value at screening of >1ng/mL
   * Soft tissue progression on CT or MRI based on RECIST 1.1 criteria or progression of bone disease according to PCWG3 criteria
9. Patients worst pain in the last 24 hours must rank less than 4 on a 0-10 scale and patients cannot be on daily narcotic medications to treat cancer-related pain. This assessment must occur within the screening window and be documented in the patient's medical record.
10. Acceptable Clinical laboratory values at Screening Visit which include:

    * Absolute neutrophil count ≥ 1000/uL; platelet count ≥ 100,000/uL, hemoglobin ≥ 8g/dL
    * Total bilirubin ≤ 1.5xULN (unless documented Gilbert's); alanine aminotransferase or aspartate aminotransferase ≤ 2.5xULN
    * Creatinine ≤ 2mg/dL
    * Hemoglobin ≤ 17.5 g/dL
11. Evidence of metastatic disease at any time point on axial imaging or bone scan, or previous biopsy. Stage IV pelvic lymph node involvement is acceptable
12. Must use a condom if having sex with a pregnant woman
13. A male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration
14. Patients may have received any number of lines of therapy for castration resistant disease

Exclusion Criteria:

1. Requires urinary catheterization for voiding due to obstruction secondary to prostatic enlargement that is well documented to be due to prostate cancer or benign prostatic hyperplasia
2. Evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone due to a potential tumor flare (e.g. high-risk bone lesions which may result in fracture or spinal cord compression
3. Clinically significant cardiovascular disease as evidenced by any of the following:

   * Myocardial infarction with 6 months of screening
   * uncontrolled angina within 3 months of screening
   * NYHA class 3 or 4 congestive heart failure
   * clinically significant ventricular arrhythmia
   * Mobitz II/Second degree/or 3rd degree heart block without a pacemaker in place; uncontrolled HTN (systolic >180mmHg or diastolic >105mmHg at screening
4. Previous exposure to a second-generation anti-androgen i.e enzalutamide or apalutamide
5. Received investigational agent within 2 weeks of screening
6. Therapy with antineoplastic systemic chemotherapy or biological therapy within 2 weeks of screening
7. Radiation therapy within 2 weeks of screening
8. History of a prior malignancy (excluding an adequately treated basal or squamous cell skin cancer, superficial bladder cancer, or a cancer in situ) within 5 years prior to study enrollment
9. History of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agent
10. Known or suspected brain metastasis or active leptomeningeal disease
11. History of seizure at any time in the past. Also, history of loss of consciousness or transient ischemic attack within 12 months of Day 1 visit
12. Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Administration of Transdermal Testosterone Alternating with Enzalutamide | Study start date to study end date, up to 12 months, or until patient death
  This study will be considered feasible if at least 50% of patients approached for participation enroll and if at least 50% of patients that initiate therapy do not withdraw consent for participation.

SECONDARY OUTCOMES:
Safety of the Administration of Transdermal Testosterone Alternating with Enzalutamide | Study start date to study end date, up to 12 months, or until patient death
  Safety will be assessed based on the Common Terminology Criteria of Adverse Events (CTCAE) v5.0 criteria, in which rates of Grade 1-5 AE will be assessed, with a prticular attention to grade 3-5 events
Prostate Specific Antigen (PSA) Response Rate | Study start date to study end date, up to 12 months, or until patient death
  PSA response rates as measured by serum PSA at designated study visits. Response will be defined as a decline in the serum PSA of 50% from baseline value at start of study.
Time to Radiographic Progression | Study start date to study end date, up to 12 months, or until patient death
  Time to radiographic progression as measured by Response Evaluation Criteria in Solid Tumors (RECIST).
Time to Radiographic Progression | Study start date to study end date, up to 12 months, or until patient death
  Time to radiographic progression as measured by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) imaging criteria.
Time to PSA Progression | Study start date to study end date, every four weeks, up to 12 months, or until patient death
  This will be defined by the PCWG3.
Maximum Decrease in PSA | Study start date to study end date, up to 12 months, or until patient death
  PSA will be assessed at baseline and every four weeks. Maximum decrease assessed through these measurements.
Physical Function Change | Study start date to study end date, up to 12 months, or until patient death
  Assessed through handgrip exercises.
Physical Function Change | Study start date to study end date, up to 12 months, or until patient death
  Assessed through chair rise exercises.
Patient Activation | Study start date to study end date, up to 12 months, or until patient death
  Assessed using the Self-Efficacy for Physical Activity Scale (SEPA), which uses a 5 point Likert scale.
Reported Fatigue | Study start date to study end date, up to 12 months, or until patient death
  Measured by the Functional Assessment of Cancer Therapy-Fatigue (FACT-Fatigue 13).
Patient Mood and Depression Evaluation | Study start date to study end date, up to 12 months, or until patient death
  Measured through the Center for Epidemiologic Studies-Depression Scale (CES-D), which uses a point system based on responses ranging from "not at all" to "all the time."
Bone Health | Study start date to study end date, up to 12 months, or until patient death
  Standard bone densometry assessment will be used to calculate T and Z score to determine normal, osteopenic, or osteoporotic bone mineral density.
Body Composition | Study start date to study end date, up to 12 months, or until patient death
  Measured by a DXA scanner. Free fat mass and lean body mass will be assessed to determine sarcopenic obesity.
Quality of Life Assessment | Study start date to study end date, up to 12 months, or until patient death
  Measured by the Functional Assessment of Cancer Therapy-Prostate (FACT-P).
Change in Hormones | Study start date to study end date, up to 12 months, or until patient death
  Change in testosterone, estrogen, and sex hormone binding globulin.
Self-Reported Physical Function | Study start date to study end date, up to 12 months, or until patient death
  Measured by the PROMIS-PA.
Energy Expenditure | Study start date to study end date, up to 12 months, or until patient death
  Measured by hood assessment.
Change in Max Repetition | Study start date to study end date, up to 12 months, or until patient death
  Measured by subject's maximal leg press over time in the energy-balance laboratory.
Change in Spontaneous Physical Activity and Sedentary Time | Study start date to study end date, up to 12 months, or until patient death
  Measured through accelerometry. Patients will wear an accelerometer for one week at initiation and again one month later.
PSA Response in this Cohort of Patients vs Historical Cohorts | Study start date to study end date, up to 12 months, or until patient death
  Assessed through IM testosterone historical data.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Graham, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The deidentified participant data will be shared after any study publication (between 6 and 36 months post publication). Study protocol also available.
Supporting Information: Study Protocol
Time Frame: Between 6 and 36 months post publication
Access Criteria: Sound proposal with IRB approval. Analyses can be be in keeping with the submitted protocol. This will be reviewed internally for use.